CLINICAL TRIAL: NCT06662448
Title: An Open-Label Study to Evaluate the Efficacy and Feasibility of Home-Based Repetitive Transorbital Alternating Current Stimulation for Optic Neuropathies
Brief Title: Repetitive Transorbital Alternating Current Stimulation for Optic Neuropathies
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-01043
Record Dates: First submitted 2024-10-25; First posted 2024-10-29 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Optic Neuropathy
MeSH Terms: conditions — Optic Nerve Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Home-based Repetitive Transorbital Alternating Current Stimulation (rtACS) (Experimental): Participants will undergo 30 stimulation sessions. The first two sessions will be administered in the office, the first one the day after the subjects' baseline visit and the second one 48 hours after the first intervention. Then subjects will conduct 28 at-home intervention sessions taking place every other day over the course of 8 weeks.
  Interventions: Device: SAVIR Alpha Synch mobile (SASm)

INTERVENTIONS:
Device: SAVIR Alpha Synch mobile (SASm) — The SAVIR Alpha Synch mobile is a device first used in office and then intended to be used for the home therapy of the visual system with non-invasive electrical stimulation.

SUMMARY:
The purpose of this study is to test the efficacy and feasibility of an intervention protocol for home-based repetitive transorbital alternating current stimulation (rtACS) for the treatment of visual impairment in people with optic neuropathy. The primary aims are to evaluate the effectiveness of home-based rtACS to ameliorate the progressive effects of vision loss functionally in the eye and the visual pathway, and in regard to people's independence (i.e., functional ability).

ELIGIBILITY:
Inclusion Criteria:

1. Age equal to or over 18 years old
2. Must have a permanent residence
3. Diagnosis of optic neuropathy
4. VF defects present in at least one eye (MD ≤ -3.00 dB) FL, FP, FN <33%
5. Visual Field Index (VFI) 10-90%
6. Clear optical apparatus
7. Best-corrected VA of 20/400 or better in at least one eye
8. Commitment to comply with study procedures: 8-week period of intervention sessions (30 sessions every other day), baseline visit, post-intervention visit, and 2 follow-up visits (2 days per visit).

   1. Scheduling
   2. Testing
9. A subject deemed incapable of performing the study intervention independently due to visual impairment or any other condition that may prevent them from performing the intervention accurately require a family member or caregiver to assist in performing the intervention.

Exclusion Criteria:

1. High intraocular pressure (over 27 mmHg)
2. End-stage organ disease or medical condition with subsequent vision loss (e.g., diabetes, stroke)
3. Advanced or unstable retinal diseases
4. Pathological nystagmus
5. Acute conjunctivitis
6. Photosensitivity to flickering lights
7. Non-ocular/ocular surgery within the previous 2 months to enrollment date
8. Electric or electronic implants (e.g., cardiac pacemaker)
9. Metallic artifacts/implants in head and/or torso (titanium screw and dental implants are allowed)
10. Diagnosed epilepsy on medical treatment
11. Auto-immune disease, acute stage (e.g., rheumatoid arthritis)
12. Metastatic disease
13. Certain mental diseases/psychiatric conditions (e.g., schizophrenia) that would affect the subject's ability to perform all necessary study tasks
14. Any chronic unstable medical conditions (e.g., uncontrolled diabetes,) that may cause a subject to miss one or more of the interventions and visits
15. Addiction (e.g., drug/alcohol dependence) that has not been in abstinent control for at least one year
16. Uncontrolled systemic hypertension (historical BP > 160/100 mmHg)
17. Pregnant or breast-feeding women or women that are planning to become pregnant, as this device has not been tested on pregnant women and there is no data on using rtACS for this particular group
18. Any severe skin condition (e.g., blisters, open wounds, cuts or irritation) or other skin defect which compromise the integrity of the skin at or near stimulation locations
19. IOP that the principal investigator determines that is not clinically stable
20. Complete blindness of both eyes
21. Non-resected brain tumors
22. Unstable diabetic retinopathy in the study eye
23. Optic neuropathies secondary to brain tumors
24. Subjects without the capacity to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2029-05-18 (Estimated); Study Completion 2029-05-18 (Estimated)

PRIMARY OUTCOMES:
Change in peripapillary retinal nerve fiber layer (RNFL) thickness (µm) | baseline, 1 week post-intervention
  Outcome measure will be assessed using Optical coherence tomography (OCT).
Change in peripapillary retinal nerve fiber layer (RNFL) thickness (µm) | baseline, 3 months post-intervention
  Outcome measure will be assessed using Optical coherence tomography (OCT).
Change in peripapillary retinal nerve fiber layer (RNFL) thickness (µm) | baseline, 6 months post-intervention
  Outcome measure will be assessed using Optical coherence tomography (OCT).
Change in macular ganglion cell-inner plexiform layer thickness (µm) | baseline, 1 week post-intervention
  Outcome measure will be assessed using Optical coherence tomography (OCT).
Change in macular ganglion cell-inner plexiform layer thickness (µm) | baseline, 3 months post-intervention
  Outcome measure will be assessed using Optical coherence tomography (OCT).
Change in macular ganglion cell-inner plexiform layer thickness (µm) | baseline, 6 months post-intervention
  Outcome measure will be assessed using Optical coherence tomography (OCT).
Change in optic nerve (ON) head cup-to-disc ratio (%) | baseline, 1 week post-intervention
  Outcome measure will be assessed using Optical coherence tomography (OCT).
Change in optic nerve (ON) head cup-to-disc ratio (%) | baseline, 3 months post-intervention
  Outcome measure will be assessed using Optical coherence tomography (OCT).
Change in optic nerve (ON) head cup-to-disc ratio (%) | baseline, 6 months post-intervention
  Outcome measure will be assessed using Optical coherence tomography (OCT).
Change in Humphrey Visual Field Analyzer (HFA) score | baseline, 1 week post-intervention
  The Humphrey Visual Field Analyzer (HFA) score is a numerical value that represents a patient's retinal sensitivity at specific points in the retina. The score is measured in decibels (dB), with higher numbers indicating higher sensitivity. A normal reading is around 30 dB, and values below this range may indicate a visual field defect. The dBs tested by the Humphrey analyzer range between 0 and 50 dB (0 is the brightest and 50 is the dimmest). A value of 0 means the patient could not see the brightest target, and a 50 means the dimmest target was seen.
Change in Humphrey Visual Field Analyzer (HFA) score | baseline, 3 months post-intervention
  The Humphrey Visual Field Analyzer (HFA) score is a numerical value that represents a patient's retinal sensitivity at specific points in the retina. The score is measured in decibels (dB), with higher numbers indicating higher sensitivity. A normal reading is around 30 dB, and values below this range may indicate a visual field defect. The dBs tested by the Humphrey analyzer range between 0 and 50 dB (0 is the brightest and 50 is the dimmest). A value of 0 means the patient could not see the brightest target, and a 50 means the dimmest target was seen.
Change in Humphrey Visual Field Analyzer (HFA) score | baseline, 6 months post-intervention
  The Humphrey Visual Field Analyzer (HFA) score is a numerical value that represents a patient's retinal sensitivity at specific points in the retina. The score is measured in decibels (dB), with higher numbers indicating higher sensitivity. A normal reading is around 30 dB, and values below this range may indicate a visual field defect. The dBs tested by the Humphrey analyzer range between 0 and 50 dB (0 is the brightest and 50 is the dimmest). A value of 0 means the patient could not see the brightest target, and a 50 means the dimmest target was seen.
Change in Early Treatment Diabetic Retinopathy Study (ETDRS) Visual Acuity (VA) score | baseline, 1 week post-intervention
  The ETDRS VA score is based on the number of letters a patient can correctly read on an ETDRS chart from a distance of 4 meters. The final score is calculated by adding 30 to the total number of letters read correctly at 4 meters.Good VA is 20/20 to 20/50; intermediate VA is <20/50 to 20/200; poor VA is <20/200.
Change in Early Treatment Diabetic Retinopathy Study (ETDRS) Visual Acuity (VA) score | baseline, 3 months post-intervention
  The ETDRS VA score is based on the number of letters a patient can correctly read on an ETDRS chart from a distance of 4 meters. The final score is calculated by adding 30 to the total number of letters read correctly at 4 meters.Good VA is 20/20 to 20/50; intermediate VA is <20/50 to 20/200; poor VA is <20/200.
Change in Early Treatment Diabetic Retinopathy Study (ETDRS) Visual Acuity (VA) score | baseline, 6 months post-intervention
  The ETDRS VA score is based on the number of letters a patient can correctly read on an ETDRS chart from a distance of 4 meters. The final score is calculated by adding 30 to the total number of letters read correctly at 4 meters.Good VA is 20/20 to 20/50; intermediate VA is <20/50 to 20/200; poor VA is <20/200.
Change in Pelli-Robson score | baseline, 1 week post-intervention
  The Pelli-Robson test is a wall-mounted chart with large letters arranged in triplets. The contrast decreases by 0.15 log units for each triplet. Patients are given credit for a contrast level if they answer two of the three letters in a triplet correctly. Each letter correctly identified is scored as 0.05 log units. The Pelli-Robson contrast sensitivity chart score range is 0.00-2.25 log contrast sensitivity. A score of 2.0 indicates normal contrast sensitivity, less than 1.5 indicates moderate reduction in contrast sensitivity, indicating some level of visual impairment, and less than 1.0 indicates visual disability.
Change in Pelli-Robson score | baseline, 3 months post-intervention
  The Pelli-Robson test is a wall-mounted chart with large letters arranged in triplets. The contrast decreases by 0.15 log units for each triplet. Patients are given credit for a contrast level if they answer two of the three letters in a triplet correctly. Each letter correctly identified is scored as 0.05 log units. The Pelli-Robson contrast sensitivity chart score range is 0.00-2.25 log contrast sensitivity. A score of 2.0 indicates normal contrast sensitivity, less than 1.5 indicates moderate reduction in contrast sensitivity, indicating some level of visual impairment, and less than 1.0 indicates visual disability.
Change in Pelli-Robson score | baseline, 6 months post-intervention
  The Pelli-Robson test is a wall-mounted chart with large letters arranged in triplets. The contrast decreases by 0.15 log units for each triplet. Patients are given credit for a contrast level if they answer two of the three letters in a triplet correctly. Each letter correctly identified is scored as 0.05 log units. The Pelli-Robson contrast sensitivity chart score range is 0.00-2.25 log contrast sensitivity. A score of 2.0 indicates normal contrast sensitivity, less than 1.5 indicates moderate reduction in contrast sensitivity, indicating some level of visual impairment, and less than 1.0 indicates visual disability.
Change in National Eye Institute Visual Functioning Questionnaire (VFQ-39) score | baseline, 1 week post-intervention
  The 39-item VFQ is designed to measure vision-related quality of life (VRQoL). It is a frequently used measure of VRQoL in vision science research. The VFQ-39 is divided into 12 subscales: general health, general vision, ocular pain, near vision, distant vision, vision specific social functioning, vision-specific role difficulties, vision-specific mental health, vision-specific dependency, driving, peripheral vision, and color vision. Responses are rated on either Likert or dichotomous (yes/no) scales. The questionnaire is scored by converting the original numeric values from the survey to a 0 to 100 scale, with 100 being the best score and 0 being the worst.
Change in National Eye Institute Visual Functioning Questionnaire (VFQ-39) score | baseline, 3 months post-intervention
  The 39-item VFQ is designed to measure VRQoL. It is a frequently used measure of VRQoL in vision science research. The VFQ-39 is divided into 12 subscales: general health, general vision, ocular pain, near vision, distant vision, vision specific social functioning, vision-specific role difficulties, vision-specific mental health, vision-specific dependency, driving, peripheral vision, and color vision. Responses are rated on either Likert or dichotomous (yes/no) scales. The questionnaire is scored by converting the original numeric values from the survey to a 0 to 100 scale, with 100 being the best score and 0 being the worst.
Change in National Eye Institute Visual Functioning Questionnaire (VFQ-39) score | baseline, 6 months post-intervention
  The 39-item VFQ is designed to measure VRQoL. It is a frequently used measure of VRQoL in vision science research. The VFQ-39 is divided into 12 subscales: general health, general vision, ocular pain, near vision, distant vision, vision specific social functioning, vision-specific role difficulties, vision-specific mental health, vision-specific dependency, driving, peripheral vision, and color vision. Responses are rated on either Likert or dichotomous (yes/no) scales. The questionnaire is scored by converting the original numeric values from the survey to a 0 to 100 scale, with 100 being the best score and 0 being the worst.

SECONDARY OUTCOMES:
Number of scheduled clinical appointments reviewed | Month 6
Number of patients considered potentially eligible as determined during review of the clinical appointment schedule | Month 6
Number of patients who are potentially eligible but express no interest in participating in the study | Month 6
Number of patients who are determined ineligible following screening procedures | Month 6
Number of participants' who adhered to the study protocol regimen | Month 6

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Panarelli, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset will be shared upon reasonable request beginning 9 to 36 months after publication or as required by a condition of awards or supporting agreements, provided the requesting investigator executes a data use agreement with NYU Langone Health. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's Data Sharing Strategy Board (DSSB). Requests should be directed to: Joseph.Panarelli@nyulangone.org. The protocol and statistical analysis plan will be posted on Clinicaltrials.gov only as required by federal regulation or supporting awards and agreements.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be provided access upon reasonable request. Requests should be directed to Joseph.Panarelli@nyulangone.org. To gain access, data requestors will need to sign a data access agreement. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's DSSB.